CLINICAL TRIAL: NCT01994291
Title: A Phase 2, Randomized, Double-Masked, Placebo-Controlled, Parallel Group, Multi-Center Study To Compare The Efficacy And Safety Of A Chemokine CCR2/5 Receptor Antagonist (PF-04634817) With That Of Ranibizumab In Adult Subjects With Diabetic Macular Edema
Brief Title: A Phase 2, Multi-Center Study To Compare The Efficacy And Safety Of A Chemokine CCR2/5 Receptor Antagonist With Ranibizumab In Adults With Diabetic Macular Edema
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1261009; 2013-003147-27 (EudraCT Number)
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Macular Edema, Diabetic
Keywords: Chemokine Antagonist; Diabetic Macular Edema; Diabetes; Diabetes Mellitus; Macular Edema; Diabetic Retinopathy; Anti-VEGF
MeSH Terms: conditions — Macular Edema; Diabetes Mellitus; Diabetic Retinopathy | interventions — Ranibizumab; PF-04634817

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Intravitreal administration of ranibizumab (either 0.3 or 0.5 mg, given monthly, as detailed in the prescribing information and label content approved for the country governing the study site) plus an oral placebo.
  Interventions: Drug: Ranibizumab; Drug: Placebo
- Arm 2 (Experimental): Oral PF-04634817 200 mg, once daily plus a masked sham therapy (given monthly).
  Interventions: Drug: PF-04634817; Drug: Masked Sham Therapy

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal Injection supplied as:
  * 10 mg/mL in a 0.2 mL vial with instructions on preparation and administration of the 0.5 mg (0.05 mL) dose.
  * 6 mg/mL in a single use vial with instructions on preparation and administration of the 0.3 mg (0.05 mL) dose.
  * Adminstered once a month for 12 weeks
  Arms: Arm 1
Drug: Placebo — Oral Placebo is provided in tablet form to match the 50mg dose of PF-04634817.
  Dose is 4 tablets each day for 12 weeks
  Arms: Arm 1
Drug: PF-04634817 — Four 50mg tablets PF-04634817 once a day for 12 weeks.
  Arms: Arm 2
Drug: Masked Sham Therapy — Empty, needle-less syringe is used by the unmasked team once a month.
  Arms: Arm 2

SUMMARY:
The study hypothesis under test is that administration of the CCR2/5 antagonist has the potential to be as effective as the current treatment options for subjects with diabetic macular edema. The current treatment option for these subjects is an injection directly into the eye, while this CCR2/5 antagonist would be an oral drug which has the potential to be just as effective. This CCR2/5 antagonist also has a broader anti-inflammatory potential and might be able to provide an alternative mechanism to treat Diabetic Macular Edema.

DETAILED DESCRIPTION:
Study recruitment was stopped on April 9, 2015. This decision was taken for business reasons due to changes in the prioritization of the drug development portfolio. This decision was not as a result of any evolving safety, efficacy issue or changes in the risk:benefit assessment of this product or regulatory interactions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diabetes Mellitus (Type 1 or Type 2) Showing Diabetic Macular Edema in the Eye
* Reduced visual acuity resulting from retinal thickening
* Female subjects of non-childbearing potential ≥18 years and male subjects greater than or equal to 18 years. A subject is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active.
* Female subjects who are not of childbearing potential must meet at least one of the following criteria:

  * Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  * Have medically confirmed ovarian failure; or
  * Achieved post-menopausal status, defined as: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal females.

Exclusion Criteria:

* Severe Impaired Renal Function
* Any intraocular condition or previous surgery in either eye that would likely require medical or surgical intervention during the study duration or if allowed to progress untreated for the 16 weeks of study duration, would likely contribute to a reduction in visual acuity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2013-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (63):
- United States (33):
  - Retina Research Institute, LLC, Phoenix, Arizona
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Sunny View Medical Center, Phoenix, Arizona
  - Premier Research Group Limited, Phoenix, Arizona
  - Retina Centers, P.C., Tucson, Arizona
  - Retina Institute of California, Arcadia, California
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Diagnostic Center, Campbell, California
  - Retina Associates of Orange County, Laguna Hills, California
  - Southern California Desert Retina Consultants, Palm Desert, California
  - American Institute of Research (Administrative Only), Whittier, California
  - New England Retina Associates, New London, Connecticut
  - Bascom Palmer Eye Institute, Miami, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - Midwest Eye Institute, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - TLC Eyecare & Laser Center, Jackson, Michigan
  - Wm Beaumont Medical Office Building, Royal Oak, Michigan
  - Charlotte Eye Ear Nose and Throat Associates PA, Charlotte, North Carolina
  - Retina Associates of Cleveland, Inc., Cleveland, Ohio
  - Retina Associates of Cleveland, Youngstown, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - University of Oklahoma -OU Physicians, Oklahoma City, Oklahoma
  - Retina Vitreous Consultants, Pittsburgh, Pennsylvania
  - Associates in Ophthalmology Ltd, West Mifflin, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Brain B.Berger,MD,PA, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
- MC Comac Medical, Sofia, Bulgaria
- Czechia (6):
  - Fakultní nemocnice Hradec Králové, Ocni klinika, Hradec Králové
  - Fakultní nemocnice Hradec Králové, Nemocnicni lekarna, Hradec Králové
  - Fakultni nemocnice Ostrava, lekarna, Ostrava - Poruba
  - Fakultni nemocnice Ostrava, Ocni klinika, Ostrava - Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Oftalmologicka klinika, Prague
  - Fakultni nemocnice Kralovske Vinohrady, Ustavni lekarna, Prague
- Germany (8):
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Universitaetsklinikum Muenster, Münster, Germany
  - Charite - Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Universitaetsmedizin Goettingen, Göttingen
  - Universitatsmedizin Mainz, Mainz
  - Augenärzte am St. Franziskus-Hospital, Münster
  - Knappschaftsklinikum GmbH, Sulzbach
  - Universitatsklinikum Tubingen, Tübingen
- Hungary (6):
  - Semmelweis Egyetem, Szemészeti Klinika, Budapest
  - Bajcsy-Zsilinszky Korhaz, Szemeszet, Budapest
  - Budapest Retina Associates Kft., Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Szemklinika, Debrecen
  - Ganglion Orvosi Kozpont, Pécs
  - Csolnoky Ferenc Korhaz, Szemeszeti Osztaly, Veszprém
- Israel (5):
  - Hadassah Medical Organization, Hadassah Medical Center, Ein Karem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Spitalul Clinic Republican, Chisinau, Moldova
- Uniwersytecki Szpital Kliniczny Im. Jana Mikulicza Radeckiego We Wrocławiu, Klinika Okulistyki, Wroclaw, Poland
- Romania (2):
  - Med Life SA, Sectia Oftalmologie, Bucharest
  - Institutul National de Diabet, Nutritie si Boli Metabolice "N.C.Paulescu", Bucharest

REFERENCES:
- [Derived] Gale JD, Berger B, Gilbert S, Popa S, Sultan MB, Schachar RA, Girgenti D, Perros-Huguet C. A CCR2/5 Inhibitor, PF-04634817, Is Inferior to Monthly Ranibizumab in the Treatment of Diabetic Macular Edema. Invest Ophthalmol Vis Sci. 2018 May 1;59(6):2659-2669. doi: 10.1167/iovs.17-22731. PMID 29847672
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1261009&StudyName=A%20Phase%202%2C%20Multi-Center%20Study%20To%20Compare%20The%20Efficacy%20And%20Safety%20Of%20A%20Chemokine%20CCR2/5%20Receptor%20Antagonist%20With%20Ranibizumab%20In%20Adult

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 199 participants were randomized, with 99 randomized to receive PF 04634817 200 mg and 99 to placebo + ranibizumab 0.3/0.5 mg. One participant was randomized but discontinued prior to dosing as no longer willing to participate.
Groups:
- PF-04634817 200 mg QD: Participants received 50 mg tablets of PF-04634817 and masked sham therapy.
- Placebo QD + Ranibizumab 0.3 mg: Participants received Ranibizumab 0.3 mg intravitreal injection and matching placebo.
- Placebo QD + Ranibizumab 0.5 mg: Participants received Ranibizumab 0.5 mg intravitreal injection and matching placebo.
Period: Overall Study
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg
Started | 99 | 43 | 56
Received Treatment | 99 | 43 | 56
Completed | 84 | 36 | 47
Not Completed | 15 | 7 | 9
Not completed — Adverse Event | 4 | 1 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Does not meet entrance criteria | 1 | 0 | 0
Not completed — Medication error without associated AE | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 3 | 5
Not completed — Other | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Total
Number analyzed (Participants) | 99 | 43 | 56 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (8.8) | 60.4 (7.5) | 63.4 (8.4) | 62.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 17 | 18 | 75
  Male | 59 | 26 | 38 | 123

OUTCOME MEASURES:

1. Primary Outcome: Mean Letter Change From Baseline at Week 12 in Best Corrected Visual Acuity (BCVA)
Description: Refraction and visual acuity were assessed through the BCVA obtained using the retro illuminated early treatment diabetic retinopathy study (ETDRS) charts. Distance visual acuity was expressed as an ETDRS score (number of letters correctly read).
Time Frame: Baseline (Day 0) and Week 12
Population: all subjects randomized and who had received at least one dose of randomized treatment and had at least one post-baseline measurement of BCVA.
Measure: Least Squares Mean (80% Confidence Interval); unit: Letters
Groups:
- Placebo QD + Ranibizumab 0.3 mg/0.5 mg: Participants received Ranibizumab 0.3 mg/0.5 mg intravitreal injection and matching placebo.
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Placebo QD + Ranibizumab 0.3 mg/0.5 mg
Number analyzed (Participants) | 87 | 38 | 53 | 91
Letters | 1.55 [-2.21 to 5.30] | 3.87 [0.09 to 7.65] | 4.03 [0.17 to 7.90] | 3.96 [0.28 to 7.64]
Statistical Analysis 1: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.3 mg; The null hypothesis was that the difference, in the mean change from baseline in BCVA in the PF-04634817 group,and the control group is less than or equal to -3 letters; Test type: Non-Inferiority or Equivalence — Non inferiority was to be declared if the lower limit of the confidence interval for the mean difference at Week 12 is greater than -3.0 letters; p = 0.1271, Mixed Models Analysis; Difference in LS means = -2.32, 80% CI 2-sided [-4.27 to -0.37], Standard Error of Mean 1.52
Statistical Analysis 2: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0699, Mixed Models Analysis; Difference in LS means = -2.48, 80% CI 2-sided [-4.24 to -0.73], Standard Error of Mean 1.36
Statistical Analysis 3: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.3 mg/0.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0399, Mixed Models Analysis; Difference in LS means = -2.41, 80% CI 2-sided [-3.91 to -0.91], Standard Error of Mean 1.17

2. Secondary Outcome: Proportion of Subjects Gaining 15 ETDRS Letters in BCVA From Baseline at Week 12
Description: Refraction and visual acuity were assessed through the BCVA obtained using the retro illuminated ETDRS charts. Distance visual acuity was expressed as an ETDRS score (number of letters correctly read).
Time Frame: Baseline (Day 0) and Week 12
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Placebo QD + Ranibizumab 0.3 mg/0.5 mg
Number analyzed (Participants) | 87 | 38 | 53 | 91
proportion of participants | 0.0690 [-2.21 to 5.30] | 0.2105 [0.09 to 7.65] | 0.1132 [0.17 to 7.90] | 0.1538 [0.28 to 7.64]
Statistical Analysis 1: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.3 mg; Test type: Superiority or Other; p = 0.0218, Barnard test; Risk Difference (RD) = -0.1416, 80% CI 2-sided [-0.2483 to -0.0467]
Statistical Analysis 2: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.5 mg; baseline in BCVA in the PF-04634817 group,and the control group is less than or equal to -3 letters; Test type: Superiority or Other; p = 0.4209, Barnard test; Risk Difference (RD) = -0.0442, 80% CI 2-sided [-0.1217 to 0.0261]
Statistical Analysis 3: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.3 mg/0.5 mg; Test type: Superiority or Other; p = 0.0778, Barnard test; Risk Difference (RD) = -0.0849, 80% CI 2-sided [-0.1516 to -0.0168]

3. Secondary Outcome: Mean Change From Baseline in Central Subfield Retinal Thickness in the Study Eye at Week 12
Description: A central reading center was used for the evaluation. A photographer or technician pre certified ("study certified") by the Central Reading Center ought to perform all optical coherence tomography (OCT) imaging. Use of a Spectralis or Cirrus OCT was acceptable.
Time Frame: Baseline (Day 0) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (80% Confidence Interval); unit: microns
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Placebo QD + Ranibizumab 0.3 mg/0.5 mg
Number analyzed (Participants) | 83 | 36 | 43 | 79
microns | 1.73 [-50.41 to 53.87] | -112.35 [-164.5 to -60.23] | -64.09 [-118.0 to -10.17] | -85.59 [-136.8 to -34.43]
Statistical Analysis 1: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.3 mg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Difference in LS means = 114.07, 80% CI 2-sided [88.56 to 139.59], Standard Error of Mean 19.84
Statistical Analysis 2: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.5 mg; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Difference in LS means = 65.81, 80% CI 2-sided [42.20 to 89.43], Standard Error of Mean 18.36
Statistical Analysis 3: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.3 mg/0.5 mg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Difference in LS means = 87.32, 80% CI 2-sided [67.45 to 107.19], Standard Error of Mean 15.44

4. Secondary Outcome: Mean Change From Baseline in The Area of Fluorescein Leakage in the Study Eye at Week 12
Description: Fluorescein Angiography (FA) using certified digital systems was taken by a photographer who had been pre-certified ("study-certified") by the Central Reading Center. They were evaluated by the Central Reading Center.
Time Frame: Baseline (Day 0) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (80% Confidence Interval); unit: mm^2
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Placebo QD + Ranibizumab 0.3 mg/0.5 mg
Number analyzed (Participants) | 86 | 36 | 50 | 86
mm^2 | 1.02 [-3.80 to 5.85] | -6.96 [-11.66 to -2.26] | -5.32 [-10.23 to -0.41] | -6.05 [-10.76 to -1.34]
Statistical Analysis 1: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.3 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in LS means = 7.98, 80% CI 2-sided [6.13 to 9.83], Standard Error of Mean 1.44
Statistical Analysis 2: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in LS means = 6.34, 80% CI 2-sided [4.70 to 7.98], Standard Error of Mean 1.28
Statistical Analysis 3: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.3 mg/0.5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in LS means = 7.07, 80% CI 2-sided [5.66 to 8.48], Standard Error of Mean 1.09

5. Secondary Outcome: Mean Change From Baseline in Steps of Diabetic Retinopathy Step (ETDRS Severity Scale) in the Study Eye at Week 12
Description: Stereo color fundus photographs using certified digital systems were taken by a photographer who had been pre-certified ("study certified") by the Central Reading Center. They were evaluated by the Central Reading Center.
Time Frame: Baseline (Day 0) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (80% Confidence Interval); unit: Letters
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Placebo QD + Ranibizumab 0.3 mg/0.5 mg
Number analyzed (Participants) | 82 | 36 | 44 | 80
Letters | 0.11 [-0.44 to 0.66] | -0.23 [-0.76 to 0.31] | -0.44 [-1.00 to 0.12] | -0.35 [-0.89 to 0.19]
Statistical Analysis 1: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.3 mg; Test type: Superiority or Other; p = 0.0423, ANCOVA; Difference in LS means = 0.34, 80% CI 2-sided [0.13 to 0.55], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.5 mg; Test type: Superiority or Other; p = 0.0004, ANCOVA; Difference in LS means = 0.55, 80% CI 2-sided [0.36 to 0.75], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: PF-04634817 200 mg QD vs Placebo QD + Ranibizumab 0.3 mg/0.5 mg; Test type: Superiority or Other; p = 0.0004, ANCOVA; Difference in LS means = 0.46, 80% CI 2-sided [0.30 to 0.63], Standard Error of Mean 0.13

6. Secondary Outcome: Plasma Concentration of PF-04634817 up to Week 12
Time Frame: Week 0, Week 4, Week 8, and Week 12
Population: All subjects in the full analysis set (FAS) for whom a pharmacokinetic sample was obtained and analyzed. The FAS was defined as all subjects randomized and who had received at least one dose of randomized treatment and had at least one post-baseline measurement of BCVA.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)/milliliter (mL)
Arm/Group | PF-04634817 200 mg QD
Number analyzed (Participants) | 96
nanogram (ng)/milliliter (mL)
  Week 0, Hour 2 (N = 91) | 612.5 (61)
  Week 4, Hour 0 (N = 88) | 180.0 (81)
  Week 4, Hour 2 (N = 87) | 682.0 (61)
  Week 8, Hour 0 (N = 90) | 159.9 (68)
  Week 8, Hour 2 (N = 89) | 752.0 (57)
  Week 12 (N = 86) | 285.2 (105)

7. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence without regard to causality in a participant who received study drug. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Week 0 to Week 16
Population: The Safety Analysis Set was defined as all subjects who receive at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Placebo QD + Ranibizumab 0.3 mg/0.5 mg
Number analyzed (Participants) | 99 | 43 | 56 | 99
participants
  Number of Participants with AEs | 53 | 32 | 27 | 59
  Number of Participants with SAEs | 7 | 2 | 3 | 5

8. Other Pre Specified Outcome: Number of Participants With Potentially Clinically Important Post-Baseline Vital Signs
Description: Number of participants who met the categorical summary of post-baseline criteria at any time point, defined as: supine pulse rate <40 beats per minute (bpm) or >120 bpm; supine systolic blood pressure (SBP) ≥30 millimeters of mercury (mmHg) change from baseline in same posture; supine diastolic BP (DBP) ≥20 mmHg change from baseline in same posture; supine SBP <90 mmHg; supine DBP <50 mmHg.
Time Frame: Week -5 to Week 16
Population: The Safety Analysis Set was defined as all subjects who receive at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Placebo QD + Ranibizumab 0.3 mg/0.5 mg
Number analyzed (Participants) | 99 | 42 | 55 | 97
participants
  Absolute Supine SBP <90 mm Hg | 1 | 0 | 0 | 0
  Increase from Baseline in Supine SBP >=30 mm Hg | 3 | 4 | 3 | 7
  Increase from Baseline in Supine DBP >=20 mm Hg | 2 | 2 | 2 | 4
  Decrease from Baseline in Supine SBP >=30 mm Hg | 3 | 0 | 2 | 2
  Decrease from Baseline in Supine DBP >=20 mm Hg | 2 | 0 | 0 | 0

9. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities
Description: The following laboratory parameters were analyzed for abnormalities at any time point: hematology (hemoglobin, hematocrit, red blood cell count (RBC), white blood cell count (WBC) with differential, and platelet count); blood chemistry (sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, albumin, calcium, total, direct and indirect bilirubin, gamma glutamyltransferase (GGT), alanine aminotransferase (ALT), aspartate aminotransferase (AST), lactic dehydrogenase (LDH), alkaline phosphatase, creatine phosphokinase (CPK), uric acid, amylase and lipase); follicle-stimulating hormone (FSH) (Weeks -5 to 0 only, for postmenopausal women who have been amenorrheic for at least 12 consecutive months prior to screening visit).
Time Frame: Week -5 to Week 16
Population: The Safety Analysis Set was defined as all subjects who receive at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Placebo QD + Ranibizumab 0.3 mg/0.5 mg
Number analyzed (Participants) | 99 | 42 | 55 | 97
participants | 45 | 19 | 21 | 40

10. Other Pre Specified Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Findings
Description: ECG parameters included PR interval, QRS interval, and corrected QT interval using Fridericia's formula (QTcF). Criteria for ECG changes meeting potential clinical concern included: PR interval greater than or equal to (>=)300 milliseconds (msec) or >=25% increase when baseline is greater than (>)200 msec and >=50% increase when baseline is less than or equal to (≤)200 msec; QRS interval >=200 msec or >=25% increase when baseline is greater than (>)200 msec and >=50% increase when baseline is less than or equal to (≤)200 msec; QT interval >=500 msec; and QTcF >=450 msec or >=30 msec increase. The number of participants with potentially clinically significant ECG findings at any visit were reported.
Time Frame: Week -5 to Week 16
Population: The Safety Analysis Set was defined as all subjects who receive at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Placebo QD + Ranibizumab 0.3 mg/0.5 mg
Number analyzed (Participants) | 99 | 43 | 56 | 99
participants
  QTcF Interval 450-<480 msec | 13 | 2 | 4 | 6
  QTcF Interval 480-<500 msec | 1 | 0 | 0 | 0
  QRS Interval >=50% increase from baseline | 0 | 1 | 0 | 1
  QTcF Interval 30-<60 msec increase from baseline | 6 | 2 | 1 | 3

11. Other Pre Specified Outcome: Number of Participants With Changes in the Anterior Segment of the Study Eye at Week 12
Description: The anterior biomicroscopy exam was done undilated in order to assess whether there was any anterior segment inflammation caused either by ranibizumab or PF-04634817.
Time Frame: Week -5 to Week 16
Population: The Safety Analysis Set was defined as all subjects who receive at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Placebo QD + Ranibizumab 0.3 mg/0.5 mg
Number analyzed (Participants) | 99 | 43 | 56 | 99
participants
  Improvement of findings in Lids | 1 | 0 | 0 | 0
  New finding (NF)/worsening of findings in Lids | 1 | 0 | 0 | 0
  Improvement of findings in conjunctiva palpebrae | 0 | 0 | 0 | 0
  NF/worsening of findings in conjunctiva palpebrae | 0 | 1 | 0 | 1
  Improvement of findings in conjunctiva bulbi | 2 | 0 | 0 | 0
  NF/worsening of findings in conjunctiva bulbi | 0 | 0 | 0 | 0
  Improvement of findings in sclera | 0 | 0 | 0 | 0
  NF/worsening of findings in sclera | 0 | 0 | 0 | 0
  Improvement of findings in cornea | 1 | 0 | 0 | 0
  NF/worsening of findings in cornea | 0 | 0 | 0 | 0
  Improvement of findings in anterior chamber | 0 | 0 | 0 | 0
  NF/worsening of findings in anterior chamber | 0 | 0 | 0 | 0
  Improvement of findings in iris | 0 | 0 | 0 | 0
  NF/worsening of findings in iris | 0 | 0 | 0 | 0
  Improvement of findings in lens | 0 | 0 | 0 | 0
  NF/worsening of findings in lens | 0 | 0 | 1 | 1

12. Other Pre Specified Outcome: Maximum Increase of Intraocular Pressure (IOP) From Baseline in Study Eye
Description: IOP was measured using Goldmann applanation tonometry. To maintain consistency, it was recommended that the same examiner ought to measure IOP with the same tonometer at each visit for a given subject. Intraocular pressure ought to be measured in the study eye approximately 30 minutes after intravitreal injection or masked sham therapy (performed by unmasked study team member).
Time Frame: Week -5 to Week 16
Population: The Safety Analysis Set was defined as all subjects who receive at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Placebo QD + Ranibizumab 0.3 mg/0.5 mg
Number analyzed (Participants) | 99 | 43 | 56 | 99
mmHg | 2.5 (2.58) | 6.0 (4.74) | 3.0 (3.32) | 4.3 (4.24)

13. Other Pre Specified Outcome: Number of Participants With Change in Ophthalmoscopy Examination Results in Study Eye After Administration of Ranibizumab or Masked Sham Therapy at Week 8
Description: Ophthalmoscopy ought to be performed after pupillary dilation to examine the vitreous body, optic nerve head, macular and peripheral retina. All findings, including the presence or absence of vitreous inflammation, ought to be documented. All post-dose ophthalmoscopy assessments ought to be made immediately following the administration of ranibizumab or masked sham therapy.
Time Frame: Week -5 to Week 16
Population: The Safety Analysis Set was defined as all subjects who receive at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg | Placebo QD + Ranibizumab 0.3 mg/0.5 mg
Number analyzed (Participants) | 99 | 43 | 56 | 99
participants
  Improvement of findings in vitreous body | 0 | 0 | 0 | 0
  NF/worsening of findings in vitreous body | 0 | 0 | 0 | 0
  Improvement of findings in optic nerve head | 0 | 0 | 0 | 0
  NF/worsening of findings in optic nerve head | 0 | 0 | 0 | 0
  Improvement of findings in retina macula | 0 | 0 | 0 | 0
  NF/worsening of findings in retina macula | 0 | 0 | 0 | 0
  Improvement of findings in retina non-macula | 0 | 0 | 0 | 0
  NF/worsening of findings in retina non-macula | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 12
Arm/Group | PF-04634817 200 mg QD | Placebo QD + Ranibizumab 0.3 mg | Placebo QD + Ranibizumab 0.5 mg
Serious Adverse Events (participants affected / at risk) | 7/99 | 2/43 | 3/56
Other Adverse Events (participants affected / at risk) | 17/99 | 15/43 | 7/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04634817 200 mg QD (N=99) | Placebo QD + Ranibizumab 0.3 mg (N=43) | Placebo QD + Ranibizumab 0.5 mg (N=56)
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Personality disorder (Psychiatric disorders) | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04634817 200 mg QD (N=99) | Placebo QD + Ranibizumab 0.3 mg (N=43) | Placebo QD + Ranibizumab 0.5 mg (N=56)
Blepharitis (Eye disorders) | 1 | 3 | 0
Conjunctival haemorrhage (Eye disorders) | 5 | 1 | 0
Diabetic retinal oedema (Eye disorders) | 4 | 7 | 3
Eye irritation (Eye disorders) | 6 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 3 | 0
Vitreous haemorrhage (Eye disorders) | 2 | 3 | 1
Intraocular pressure increased (Investigations) | 0 | 1 | 3
Headache (Nervous system disorders) | 3 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.